CLINICAL TRIAL: NCT00494923
Title: Glaucoma Including Pseudoexfoliation Syndrome (SFB 539)
Brief Title: Early Diagnosis, Pathogenesis and Progression of Open Angle Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: DFG-SFB539-R
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Primary Open Angle Glaucoma; Secondary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The Erlangen Glaucoma Registry is a clinical registry for cross sectional and longitudinal observation of patients with open angle glaucoma (OAG) or glaucoma suspect, founded in 1991. The primary aim is the evaluation of diagnostic and prognostic validity of morphometrical, sensory and hemodynamical diagnostic procedures. No therapeutic studies are performed.

DETAILED DESCRIPTION:
Purpose: Detection of onset and progression of structural and functional damage due to glaucoma. Determination of rate and amount of progressive change due to glaucoma. Characterisation of the relationship between structural and functional change over time. Evaluation of predictive factors for the development and progression of glaucoma.

ELIGIBILITY:
Participants:

* Patients: Primary open angle glaucoma, secondary open angle glaucoma due to PEX or MDS, glaucoma suspects including ocular hypertension
* Healthy volunteers (for cross sectional analysis only)

Inclusion Criteria:

* Open anterior chamber angle
* Best corrected visual acuity 0.7 or better
* Age between 18 and 65 years

Exclusion Criteria:

* Any eye disease other than glaucoma
* Systemic diseases with potentially ocular involvement (e.g., diabetes mellitus)
* Myopic or hyperopic refractive error exceeding 8.0 diopters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 1999-01; Primary Completion 2015-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression | up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Anselm G Juenemann, Prof., Study Chair — University Erlangen-Nuremberg
Locations (1):
- University Eye Hospital, Erlangen, Germany

REFERENCES:
- [Result] Wessel JM, Horn FK, Tornow RP, Schmid M, Mardin CY, Kruse FE, Juenemann AG, Laemmer R. Longitudinal analysis of progression in glaucoma using spectral-domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 May 1;54(5):3613-20. doi: 10.1167/iovs.12-9786. PMID 23633657
- [Result] Hoesl LM, Tornow RP, Schrems WA, Horn FK, Mardin CY, Kruse FE, Juenemann AG, Laemmer R. Glaucoma diagnostic performance of GDxVCC and spectralis OCT on eyes with atypical retardation pattern. J Glaucoma. 2013 Apr-May;22(4):317-24. doi: 10.1097/IJG.0b013e318237c8c5. PMID 22027931
- [Result] Schrems WA, Laemmer R, Hoesl LM, Horn FK, Mardin CY, Kruse FE, Tornow RP. Influence of atypical retardation pattern on the peripapillary retinal nerve fibre distribution assessed by scanning laser polarimetry and optical coherence tomography. Br J Ophthalmol. 2011 Oct;95(10):1437-41. doi: 10.1136/bjo.2010.190074. Epub 2011 Jan 17. PMID 21242583
- [Result] Hoesl LM, Mardin CY, Horn FK, Juenemann AG, Laemmer R. Influence of glaucomatous damage and optic disc size on glaucoma detection by scanning laser tomography. J Glaucoma. 2009 Jun-Jul;18(5):385-9. doi: 10.1097/IJG.0b013e3181845ffd. PMID 19525729
- [Result] Schrems WA, Mardin CY, Horn FK, Juenemann AG, Laemmer R. Comparison of scanning laser polarimetry and optical coherence tomography in quantitative retinal nerve fiber assessment. J Glaucoma. 2010 Feb;19(2):83-94. doi: 10.1097/IJG.0b013e3181a2fc0e. PMID 19373100
- [Result] Horn FK, Mardin CY, Laemmer R, Baleanu D, Juenemann AM, Kruse FE, Tornow RP. Correlation between local glaucomatous visual field defects and loss of nerve fiber layer thickness measured with polarimetry and spectral domain OCT. Invest Ophthalmol Vis Sci. 2009 May;50(5):1971-7. doi: 10.1167/iovs.08-2405. Epub 2009 Jan 17. PMID 19151389
- [Result] Laemmer R, Schroeder S, Martus P, Viestenz A, Mardin CY. Quantification of neuroretinal rim loss using digital planimetry in long-term follow-up of normals and patients with ocular hypertension. J Glaucoma. 2007 Aug;16(5):430-6. doi: 10.1097/IJG.0b013e31804a5e80. PMID 17700284
- [Result] Laemmer R, Horn FK, Viestenz A, Juenemann AG, Mardin CY. Influence of optic disc size on parameters of retinal nerve fiber analysis with laser scanning polarimetry. Graefes Arch Clin Exp Ophthalmol. 2006 May;244(5):603-8. doi: 10.1007/s00417-005-0125-1. Epub 2005 Sep 21. PMID 16175374
- [Result] Tornow RP, Schrems WA, Bendschneider D, Horn FK, Mayer M, Mardin CY, Lammer R. Atypical retardation patterns in scanning laser polarimetry are associated with low peripapillary choroidal thickness. Invest Ophthalmol Vis Sci. 2011 Sep 29;52(10):7523-8. doi: 10.1167/iovs.11-7557. PMID 21862653
- [Result] Horn FK, Lammer R, Mardin CY, Junemann AG, Michelson G, Lausen B, Adler W. Combined evaluation of frequency doubling technology perimetry and scanning laser ophthalmoscopy for glaucoma detection using automated classification. J Glaucoma. 2012 Jan;21(1):27-34. doi: 10.1097/IJG.0b013e3182027766. PMID 21173705
- [Result] Pasutto F, Krumbiegel M, Mardin CY, Paoli D, Lammer R, Weber BH, Kruse FE, Schlotzer-Schrehardt U, Reis A. Association of LOXL1 common sequence variants in German and Italian patients with pseudoexfoliation syndrome and pseudoexfoliation glaucoma. Invest Ophthalmol Vis Sci. 2008 Apr;49(4):1459-63. doi: 10.1167/iovs.07-1449. PMID 18385063
- [Derived] Crux K, Huchzermeyer C, Kremers J, Horn FK. Objective detection of visual field defects with multifrequency VEPs. Doc Ophthalmol. 2024 Feb;148(1):15-24. doi: 10.1007/s10633-023-09949-4. Epub 2023 Sep 26. PMID 37749441
- [Derived] Dussan Molinos L, Huchzermeyer C, Lammer R, Kremers J, Horn FK. Blue-Yellow VEP with Projector-Stimulation in Glaucoma. Graefes Arch Clin Exp Ophthalmol. 2022 Apr;260(4):1171-1181. doi: 10.1007/s00417-021-05473-w. Epub 2021 Nov 25. PMID 34821990
- [Derived] Thiermeier N, Lammer R, Mardin C, Hohberger B. Erlanger Glaucoma Registry: Effect of a Long-Term Therapy with Statins and Acetyl Salicylic Acid on Glaucoma Conversion and Progression. Biology (Basel). 2021 Jun 16;10(6):538. doi: 10.3390/biology10060538. PMID 34208432
- [Derived] Denkel L, Hohberger B, Lammer R. Influence of Mitomycin C on the Therapeutic Success of Stand-Alone Xen45 Gel Stents and Its Combination with Cataract Surgery in Open-Angle Glaucoma Patients. Klin Monbl Augenheilkd. 2021 Aug;238(8):861-867. doi: 10.1055/a-1384-1020. Epub 2021 May 17. PMID 34000747
- [Derived] Hohberger B, Lucio M, Schlick S, Wollborn A, Hosari S, Mardin C. OCT-angiography: Regional reduced macula microcirculation in ocular hypertensive and pre-perimetric glaucoma patients. PLoS One. 2021 Feb 11;16(2):e0246469. doi: 10.1371/journal.pone.0246469. eCollection 2021. PMID 33571215
- [Derived] Tornow RP, Kolar R, Odstrcilik J, Labounkova I, Horn F. Imaging video plethysmography shows reduced signal amplitude in glaucoma patients in the area of the microvascular tissue of the optic nerve head. Graefes Arch Clin Exp Ophthalmol. 2021 Feb;259(2):483-494. doi: 10.1007/s00417-020-04934-y. Epub 2020 Sep 22. PMID 32960321
- [Derived] Hohberger B, Kunze R, Wallukat G, Kara K, Mardin CY, Lammer R, Schlotzer-Schrehardt U, Hosari S, Horn F, Munoz L, Herrmann M. Autoantibodies Activating the beta2-Adrenergic Receptor Characterize Patients With Primary and Secondary Glaucoma. Front Immunol. 2019 Oct 1;10:2112. doi: 10.3389/fimmu.2019.02112. eCollection 2019. PMID 31632387
- [Derived] Edlinger FSM, Schrems-Hoesl LM, Mardin CY, Laemmer R, Kruse FE, Schrems WA. Structural changes of macular inner retinal layers in early normal-tension and high-tension glaucoma by spectral-domain optical coherence tomography. Graefes Arch Clin Exp Ophthalmol. 2018 Jul;256(7):1245-1256. doi: 10.1007/s00417-018-3944-6. Epub 2018 Mar 9. PMID 29523993
- [Derived] Junemann A, Hohberger B, Rech J, Sheriff A, Fu Q, Schlotzer-Schrehardt U, Voll RE, Bartel S, Kalbacher H, Hoebeke J, Rejdak R, Horn F, Wallukat G, Kunze R, Herrmann M. Agonistic Autoantibodies to the beta2-Adrenergic Receptor Involved in the Pathogenesis of Open-Angle Glaucoma. Front Immunol. 2018 Feb 12;9:145. doi: 10.3389/fimmu.2018.00145. eCollection 2018. PMID 29483909
- [Derived] Schrems-Hoesl LM, Schrems WA, Laemmer R, Kruse FE, Mardin CY. Precision of Optic Nerve Head and Retinal Nerve Fiber Layer Parameter Measurements by Spectral-domain Optical Coherence Tomography. J Glaucoma. 2018 May;27(5):407-414. doi: 10.1097/IJG.0000000000000875. PMID 29329141
- [Derived] Diekmann T, Schrems-Hoesl LM, Mardin CY, Laemmer R, Horn FK, Kruse FE, Schrems WA. Predictive Factors for Visual Field Conversion: Comparison of Scanning Laser Polarimetry and Optical Coherence Tomography. J Glaucoma. 2018 Feb;27(2):157-163. doi: 10.1097/IJG.0000000000000833. PMID 29194206
- [Derived] Gmeiner JM, Schrems WA, Mardin CY, Laemmer R, Kruse FE, Schrems-Hoesl LM. Comparison of Bruch's Membrane Opening Minimum Rim Width and Peripapillary Retinal Nerve Fiber Layer Thickness in Early Glaucoma Assessment. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT575-84. doi: 10.1167/iovs.15-18906. PMID 27547890
- [Derived] Schrems-Hoesl LM, Schrems WA, Laemmer R, Horn FK, Juenemann AG, Kruse FE, Mardin CY. Confocal Laser Scanning Tomography to Predict Visual Field Conversion in Patients With Ocular Hypertension and Early Glaucoma. J Glaucoma. 2016 Apr;25(4):371-6. doi: 10.1097/IJG.0000000000000171. PMID 25304282
- [Derived] La Mancusa A, Horn FK, Kremers J, Huchzermeyer C, Rudolph M, Junemann A. Pattern electroretinograms during the cold pressor test in normals and glaucoma patients. Invest Ophthalmol Vis Sci. 2014 Apr 7;55(4):2173-9. doi: 10.1167/iovs.13-13392. PMID 24576876
- [Derived] Horn FK, Tornow RP, Junemann AG, Laemmer R, Kremers J. Perimetric measurements with flicker-defined form stimulation in comparison with conventional perimetry and retinal nerve fiber measurements. Invest Ophthalmol Vis Sci. 2014 Apr 11;55(4):2317-23. doi: 10.1167/iovs.13-12469. PMID 24355823
- [Derived] Horn FK, Kaltwasser C, Junemann AG, Kremers J, Tornow RP. Objective perimetry using a four-channel multifocal VEP system: correlation with conventional perimetry and thickness of the retinal nerve fibre layer. Br J Ophthalmol. 2012 Apr;96(4):554-9. doi: 10.1136/bjophthalmol-2011-300844. Epub 2011 Nov 24. PMID 22116959
- [Derived] Barboni MT, Pangeni G, Ventura DF, Horn F, Kremers J. Heterochromatic flicker electroretinograms reflecting luminance and cone opponent activity in glaucoma patients. Invest Ophthalmol Vis Sci. 2011 Aug 29;52(9):6757-65. doi: 10.1167/iovs.11-7538. PMID 21778269